CLINICAL TRIAL: NCT07309666
Title: Research, Development, and Application of Intelligent Diagnostic System for Orthostatic Hypotension
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: AF-SW-01-01.0
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Orthostatic Hypotension
Keywords: Orthostatic Hypotension; Blood Pressure; Cerebral Blood Flow Velocity; Cerebral Autoregulation; Risk Stratification
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OH Group: This study enrolls patients diagnosed with orthostatic hypotension (OH). Participants must have one of the following underlying conditions: 1) clinically established or probable Parkinson's disease; 2) clinically diagnosed multiple system atrophy; or 3) diabetes mellitus and aged ≥50 years. All participants in this group must meet the standard diagnostic criteria for OH (a decrease in systolic blood pressure of ≥20 mmHg or a decrease in diastolic blood pressure of ≥10 mmHg within 3 minutes of standing).
  Interventions: Other: Intelligent diagnostic system for orthostatic hypotension
- Non-OH Control Group: This study also enrolls a control group of patients without orthostatic hypotension (OH). Control participants must have the same underlying diseases as the OH group (Parkinson's disease, multiple system atrophy, or diabetes mellitus aged ≥50 years) but do not meet the diagnostic criteria for OH during the active standing test. This group is used for comparison with the OH group regarding cerebrovascular hemodynamic parameters and clinical outcomes.
  Interventions: Other: Intelligent diagnostic system for orthostatic hypotension

INTERVENTIONS:
Other: Intelligent diagnostic system for orthostatic hypotension — All participants will undergo a standardized multi-parameter monitoring protocol. After resting in the supine position for at least 10 minutes, participants will perform an active standing test. During this protocol, the following parameters are continuously and synchronously recorded using the integrated intelligent diagnostic system: non-invasive beat-to-beat blood pressure, cerebral blood flow velocity in the middle cerebral artery (assessed via transcranial Doppler, TCD), electrocardiogram (ECG), and end-tidal carbon dioxide (ETCO₂). Monitoring is conducted for a 10-minute baseline period in the supine position and continues for up to 10 minutes following standing.

SUMMARY:
Orthostatic hypotension (OH) has a high incidence rate of 30%-50% in the elderly and populations with neurodegenerative diseases. The resulting cerebral hypoperfusion significantly increases the risk of cerebral ischemia, falls, and cognitive decline. Traditional OH diagnosis primarily relies on intermittent cuff blood pressure measurements, leading to low detection rates and an inability to provide scientifically effective OH classification. Furthermore, existing research often overlooks cerebral hemodynamic mechanisms, particularly the assessment of dynamic cerebral autoregulation (dCA), making it difficult to study the mechanisms behind OH and its associated symptoms.

To address these issues, the research team has preliminarily developed an "Intelligent Diagnostic System for Orthostatic Hypotension". This system innovatively integrates synchronous and continuous monitoring of multiple parameters, including non-invasive beat-to-beat blood pressure, transcranial Doppler (TCD) cerebral blood flow velocity, and electrocardiogram (ECG). It also enables the quantitative assessment of dynamic cerebral autoregulation function. The project will collaborate with fifteen high-level clinical centers in China to collect data from 2000 patients with orthostatic hypotension. The aim is to establish and externally validate a risk stratification model for OH. By integrating multimodal clinical and hemodynamic data, the investigators intend to construct an automated, precise intelligent system for the classification, subtyping, and risk stratification of OH. This initiative will establish a standardized diagnostic and management pathway covering early screening, precise classification, early warning, and stratified intervention. The goal is to provide key technological support for enhancing the early identification and standardized management of OH, thereby reducing its associated disability and mortality rates.

DETAILED DESCRIPTION:
This prospective, multicenter, observational cohort study aims to develop and validate an intelligent diagnostic and risk stratification system for orthostatic hypotension (OH). The study plans to enroll approximately 2000 participants from 15 tertiary clinical centers in China between March 2026 and February 2029. The target population comprises adult patients (≥18 years) with Parkinson's disease (PD) or multiple system atrophy (MSA), and patients aged ≥50 years with diabetes mellitus who are suspected or diagnosed with OH. A key technical inclusion criterion is the presence of adequate bilateral temporal bone windows for reliable transcranial Doppler (TCD) monitoring.

The core methodology involves synchronous, continuous, and non-invasive monitoring of beat-to-beat blood pressure (BP), bilateral cerebral blood flow velocity (CBFv) in the middle cerebral arteries, electrocardiogram (ECG), and end-tidal carbon dioxide (PetCO₂) during a standardized active standing test. Following a 10-minute supine rest, participants rapidly stand and remain upright for up to 10 minutes. Using this integrated data stream, OH is classified as Initial, Classic, or Delayed per consensus hemodynamic thresholds. Dynamic cerebral autoregulation (dCA) is quantitatively assessed offline via transfer function analysis (TFA) of the BP and CBFv signals, deriving phase, gain (absolute and normalized), and coherence parameters in very low frequency (VLF) and low frequency (LF) bands.

Participants are followed for 24 months, with a telephone follow-up at 12 months and an in-person visit at 24 months that includes a repeat stand test and cognitive assessment. The primary technical endpoints are the algorithm-based classification of OH subtype/etiology and the quantitative dCA parameters. Secondary endpoints include the performance (sensitivity, specificity, area under the curve [AUC]) of the derived multimodal risk model in predicting clinical events such as falls, syncope, cognitive decline, and all-cause mortality.

Data analysis will involve machine learning/statistical modeling on a development cohort to generate the risk stratification model, followed by external validation on a separate cohort to assess generalizability and clinical utility.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old).
2. Clinical diagnosis of Parkinson's disease (PD) OR multiple system atrophy (MSA) OR diabetes mellitus (if diabetic, must be aged ≥50 years).
3. Suspected or diagnosed with orthostatic hypotension (OH).
4. Presence of adequate acoustic temporal bone windows for Transcranial Doppler (TCD) monitoring.
5. Willing and able to provide informed consent.

Exclusion Criteria:

1. Significant intracranial or extracranial arterial stenosis (≥70% confirmed by ultrasound).
2. Recent stroke or intracerebral hemorrhage (confirmed by CT/MRI).
3. Severe cardiac arrhythmias (e.g., atrial fibrillation) or severe valvular heart disease.
4. Bilateral temporal bone windows insufficient for TCD monitoring.
5. Pregnancy or lactation.
6. Inability to cooperate with the testing procedures.
7. Other systemic diseases that significantly affect cerebral blood flow regulation (e.g., severe thyroid or renal dysfunction).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective, multicenter study aims to enroll approximately 2000 hospitalized adult patients with Parkinson's disease, multiple system atrophy, or diabetes (aged ≥50 for diabetics) who are suspected of having or are diagnosed with orthostatic hypotension (OH). Participants will be recruited from 15 high-level clinical centers in China between March 2026 and February 2029.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Classification of Orthostatic Hypotension | 2years
  Orthostatic hypotension will be subtyped according to the timing of blood pressure reduction after standing: Classical, Initial, or Delayed. Additionally, etiology will be classified as Neurogenic or Non-neurogenic, determined by the heart rate response to blood pressure change, quantified as the ratio of change in heart rate to change in systolic blood pressure (ΔHR/ΔSBP ratio).
Dynamic Cerebral Autoregulation Parameters | 2years
  Quantitative assessment of dynamic cerebral autoregulation (dCA) function will be performed using Transfer Function Analysis (TFA) on continuous blood pressure and cerebral blood flow velocity signals. Parameters include phase difference, gain, and coherence in the following frequency ranges: very low frequency (VLF: 0.02-0.07 Hz), low frequency (LF: 0.07-0.20 Hz), and high frequency (HF: 0.20-0.70 Hz).

SECONDARY OUTCOMES:
Performance of the Risk Stratification Model | At the end of the 24-month follow-up period, when outcome data for all participants are available for model validation.
  The predictive accuracy of the developed risk stratification model for adverse events (e.g., falls, syncope) will be assessed using metrics including sensitivity, specificity, and the area under the receiver operating characteristic curve (AUC).
Incidence of Adverse Clinical Events | Assessed at 12-month and 24-month follow-up visits.
  The cumulative incidence of the following clinical events will be recorded and compared between groups: falls, syncope (fainting), fractures, cognitive decline (defined as a decrease in Montreal Cognitive Assessment [MoCA] or Mini-Mental State Examination [MMSE] score from baseline), and all-cause mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wieling W, Kaufmann H, Claydon VE, van Wijnen VK, Harms MPM, Juraschek SP, Thijs RD. Diagnosis and treatment of orthostatic hypotension. Lancet Neurol. 2022 Aug;21(8):735-746. doi: 10.1016/S1474-4422(22)00169-7. PMID 35841911
- [Background] Freeman R, Abuzinadah AR, Gibbons C, Jones P, Miglis MG, Sinn DI. Orthostatic Hypotension: JACC State-of-the-Art Review. J Am Coll Cardiol. 2018 Sep 11;72(11):1294-1309. doi: 10.1016/j.jacc.2018.05.079. PMID 30190008
- [Background] Thijs RD, Brignole M, Falup-Pecurariu C, Fanciulli A, Freeman R, Guaraldi P, Jordan J, Habek M, Hilz M, Pavy-LeTraon A, Stankovic I, Struhal W, Sutton R, Wenning G, van Dijk JG. Recommendations for tilt table testing and other provocative cardiovascular autonomic tests in conditions that may cause transient loss of consciousness : Consensus statement of the European Federation of Autonomic Societies (EFAS) endorsed by the American Autonomic Society (AAS) and the European Academy of Neurology (EAN). Auton Neurosci. 2021 Jul;233:102792. doi: 10.1016/j.autneu.2021.102792. Epub 2021 Mar 19. PMID 33752997
- [Background] Juraschek SP, Daya N, Rawlings AM, Appel LJ, Miller ER 3rd, Windham BG, Griswold ME, Heiss G, Selvin E. Association of History of Dizziness and Long-term Adverse Outcomes With Early vs Later Orthostatic Hypotension Assessment Times in Middle-aged Adults. JAMA Intern Med. 2017 Sep 1;177(9):1316-1323. doi: 10.1001/jamainternmed.2017.2937. PMID 28738139
- [Background] Panerai RB, Brassard P, Burma JS, Castro P, Claassen JA, van Lieshout JJ, Liu J, Lucas SJ, Minhas JS, Mitsis GD, Nogueira RC, Ogoh S, Payne SJ, Rickards CA, Robertson AD, Rodrigues GD, Smirl JD, Simpson DM; Cerebrovascular Research Network (CARNet). Transfer function analysis of dynamic cerebral autoregulation: A CARNet white paper 2022 update. J Cereb Blood Flow Metab. 2023 Jan;43(1):3-25. doi: 10.1177/0271678X221119760. Epub 2022 Aug 12. PMID 35962478